CLINICAL TRIAL: NCT05767034
Title: A Randomized, Parallel-group, Double-blind, Placebo-controlled, Multicenter Phase III Trial to Evaluate Efficacy and Safety of Secukinumab Administered Subcutaneously Versus Placebo, in Combination With a Glucocorticoid Taper Regimen, in Patients With Polymyalgia Rheumatica (PMR)
Brief Title: Phase III Study of Efficacy and Safety of Secukinumab Versus Placebo, in Combination With Glucocorticoid Taper Regimen, in Patients With Polymyalgia Rheumatica (PMR)
Acronym: REPLENISH
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457C22301; 2022-501895-25-00 (Other: EU CT Number)
Record Dates: First submitted 2023-03-06; First posted 2023-03-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Polymyalgia Rheumatica
Keywords: Polymyalgia Rheumatica; secukinumab; monoclonal antibody; prednisone taper regimen; glucocorticoid; PMR
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Secukinumab 300 mg (Experimental): randomized in 1:1:1 ratio every 4 weeks
  Interventions: Drug: Secukinumab 300 mg
- Secukinumab 150 mg (Experimental): randomized in 1:1:1 ratio every 4 weeks
  Interventions: Drug: Secukinumab 150 mg
- Placebo to secukinumab (Placebo Comparator): randomized in 1:1:1 ratio every 4 weeks
  Interventions: Other: Placebo to secukinumab

INTERVENTIONS:
Drug: Secukinumab 300 mg — Taken subcutaneously every 4 weeks until Week 48 in combination with a 24-week prednisone taper regimen
  Other Names: AIN457
  Arms: Secukinumab 300 mg
Drug: Secukinumab 150 mg — Taken subcutaneously every 4 weeks until Week 48 in combination with a 24-week prednisone taper regimen
  Other Names: AIN457
  Arms: Secukinumab 150 mg
Other: Placebo to secukinumab — Taken subcutaneously every 4 weeks until Week 48 in combination with a 24-week prednisone taper regimen
  Arms: Placebo to secukinumab

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of secukinumab 300 milligram (mg) and 150 mg administered subcutaneously (s.c.) for 52 weeks in combination with prednisone tapered over 24 weeks in adult participants with PMR who have recently relapsed.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel group study with two secukinumab dose regimens in approximately 360 PMR patients who had recently relapsed. The study consists of: screening (up to 6 weeks); treatment period (52 weeks, with last IMP administration at 48 weeks, active drug or placebo) in combination with prednisone tapered over 24 weeks; treatment-free follow-up (up to 24 weeks). Adult males and females of at least 50 years of age with a recent PMR relapse (within 12 weeks from Baseline) will be included. Dosing will be once every week for the first 4 weeks, and once every 4 weeks thereafter via pre-filled syringe.

The primary objective is to demonstrate the efficacy of secukinumab 300 mg subcutaneously in combination with a 24-week glucocorticoid (GC) taper regimen compared with placebo with respect to the proportion of patients in sustained remission at Week 52. Primary secondary objectives are to assess difference in proportion of patients achieving complete sustained remission at Week 52, adjusted annual cumulative GC dose and time to first use of escape treatment or rescue treatment through Week 52. Key safety data will be collected, along with Patient Reported Outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study
* Male or non-pregnant, non-lactating female participants at least 50 years of age.
* Diagnosis of PMR according to the provisional American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria: Participants ≥ 50 years of age with a history of bilateral shoulder pain accompanied by elevated C-reactive protein (CRP) concentration (≥ 10 mg/L) and/or elevated erythrocyte sedimentation rate (ESR) (≥ 30 mm/hr) who scored at least 4 points from the following optional classification criteria:

  * Morning stiffness > 45 minutes (min) (2 points)
  * Hip pain or restricted range of motion (1 point)
  * Absence of rheumatoid factor and/or anti-citrullinated protein antibodies (2 points)
  * Absence of other joint involvement (1 point)
* Participants must have a history of being treated for at least 8 consecutive weeks with prednisone ≥ 10 mg/day, or equivalent dose of another GC at any time prior to screening
* Participants must have had at least one episode of PMR relapse while attempting to taper prednisone at a dose that is ≥ 5 mg/day (or equivalent dose of another GC) within the past 12 weeks prior to BSL. Diagnosis of a PMR relapse is defined as participant meeting both of the following:

  * Recurrence of bilateral shoulder girdle and/or bilateral hip girdle pain associated with inflammatory stiffness with or without additional symptoms indicative of PMR relapse (such as constitutional symptoms) within 12 weeks prior to BSL that are in the opinion of the Investigator not due to other diseases that may mimic PMR such as osteoarthritis in shoulders or hips, polyarticular calcium pyrophosphate deposition disease, rotator cuff disease, adhesive capsulitis (frozen shoulder) or fibromyalgia.
  * Elevated ESR (≥ 30 mm/hr) and/or elevated CRP (> upper limit of normal (ULN)) attributable to PMR at the time of relapse and/or at screening
* Participants must have been treated as per local treatment recommendations following the latest PMR relapse and must be on prednisone of at least 7.5 mg/day (or equivalent) and not exceeding 25 mg/day at screening and during the screening period

Exclusion Criteria:

* Evidence/history of GCA as indicated by typical (cranial) symptoms (e.g., persistent or recurrent localized headache, temporal artery or scalp tenderness, jaw claudication, blurry or loss of vision, symptoms of stroke), extremity claudication, imaging and/or temporal artery biopsy result
* Concurrent rheumatoid arthritis or other inflammatory arthritis or other connective tissue diseases, such as but not limited to systemic lupus erythematosus, systemic sclerosis, vasculitis, myositis, mixed connective tissue disease, and ankylosing spondylitis
* Concurrent diagnosis or history of neuropathic muscular diseases or fibromyalgia
* Inadequately treated hypothyroidism (e.g., persistence of symptoms, lack of normalization of serum TSH despite regular hormonal replacement treatment)
* Previous exposure to secukinumab or other biologic drug directly targeting IL-17 or IL-17 receptor
* Participants treated with tocilizumab or other IL-6/IL6-receptor inhibitors within 12 weeks or within 5 half-lives (whichever is longer) prior to BSL; participant who did not respond to or experienced a relapse during treatment are excluded from enrollment into the study Other protocol-defined inclusion/exclusion criteria may apply

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2026-02-17 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving sustained remission | at Week 52
  Sustained remission at Week 52 is defined as a participant meeting all of the following:
  ● achieved remission at Week 12
  AND all of the following, sustained from Week 12 to Week 52:
  * no recurrence of signs or symptoms, attributable to PMR, that requires escape treatment or rescue treatment
  * no new diagnosis of Giant cell arteritis (GCA), that requires escape treatment or rescue treatment
  Remission at Week 12 is defined as a participant meeting all of the following at Week 12:
  * no use of escape treatment or rescue treatment prior to Week 12
  * no signs or symptoms attributable to PMR, that requires escape treatment or use of rescue treatment, at Week 12
  * no new diagnosis of GCA, that requires escape treatment or rescue treatment, at Week 12

SECONDARY OUTCOMES:
Proportion of patients achieving complete sustained remission | 52 Weeks
  Complete sustained remission at Week 52 is defined as participant meeting all of the following:
  * achieved sustained remission
  * no clinically relevant elevation of Erythrocyte sedimentation Rate (ESR) and/or C-reactive protein (CRP) at ≥2 consecutive scheduled visits from Week 12 to Week 52
Adjusted annual cumulative glucocorticoid (GC) dose adjusted by duration of study follow-up | 52 Weeks
  Adjusted annual cumulative GC dose is cumulative GC dose through Week 52 adjusted by duration of study follow-up
Time to first use of escape treatment or rescue treatment as measured in days | 52 Weeks
  First use of escape treatment or rescue treatment is defined as the first time when the escape treatment or rescue treatment is used
Change in FACIT-Fatigue Score | 52 Weeks
  The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function.
  The purpose of collecting available FACIT-Fatigue data is to assess the impact of fatigue on participants with PMR.
Change in HAQ-DI score | 52 Weeks
  The Health Assessment Questionnaire - Disability Index (HAQ-DI) is used to assess the long-term influence of chronic disease on a participant's level of functional ability and activity restriction. The purpose of the HAQ-DI is to assess the functional ability of subjects with PMR.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (123):
- United States (22):
  - Arizona Arthritis and Rheumatology Associates PLLC, Avondale, Arizona
  - Sun Valley Arthritis Center Ltd, Peoria, Arizona
  - AZ Arthritis and Rheumtlgy Rsh PLLC, Phoenix, Arizona
  - Precn Comprehensive Clnl Rsch Solns, San Leandro, California
  - Providence Saint Johns Health Ctr, Santa Monica, California
  - Center for Rheumatology Research, West Hills, California
  - Millennium Clinical Trials, Westlake Village, California
  - Rheumatology Associates of South Florida, Boca Raton, Florida
  - UF Health Cancer Center, Gainesville, Florida
  - Sarasota Arthritis Res Ctr, Sarasota, Florida
  - West Broward Rheumatology Associates Inc, Tamarac, Florida
  - Southeastern Rheumatology Alliance, Gainesville, Georgia
  - Klein and Associates, Hagerstown, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Clinical Research Inst of MI, Saint Clair Shores, Michigan
  - Kansas City Physician Partners, Kansas City, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Paramount Med Rsrch and Consult LLC, Middleburg Heights, Ohio
  - Prolato Clinical Research Center, Houston, Texas
  - DM Clinical Research, Houston, Texas
  - Accurate Clinical Research Inc, San Antonio, Texas
  - Advanced Rheumatology of Houston, Spring, Texas
- Argentina (3):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Australia (3):
  - Novartis Investigative Site, Parramatta, New South Wales
  - Novartis Investigative Site, Southport, Queensland
  - Novartis Investigative Site, Heidelberg Heights, Victoria
- Belgium (2):
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Brazil (3):
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, São Paulo
- Novartis Investigative Site, Québec, Quebec, Canada
- Chile (2):
  - Novartis Investigative Site, Viña del Mar, Región de Valparaíso
  - Novartis Investigative Site, Santiago, Santiago Metropolitan
- Colombia (3):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Cali, Valle del Cauca Department
- Czechia (6):
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Hlučín
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
  - Novartis Investigative Site, Zlín
- Denmark (4):
  - Novartis Investigative Site, Aarhus N
  - Novartis Investigative Site, Esbjerg
  - Novartis Investigative Site, Gandrup
  - Novartis Investigative Site, Vejle
- France (13):
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Toulon, Val De Marne
  - Novartis Investigative Site, Aix-en-Provence
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Cholet
  - Novartis Investigative Site, Colmar
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (8):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Ratingen
  - Novartis Investigative Site, Rendsburg
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Veszprém
- Novartis Investigative Site, Reykjavik, Iceland
- Novartis Investigative Site, Dublin, Ireland
- Israel (2):
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (5):
  - Novartis Investigative Site, Bolzano, BZ
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Reggio Emilia, RE
- Japan (17):
  - Novartis Investigative Site, Ichikawa, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Nagano, Nagano
  - Novartis Investigative Site, Beppu, Oita Prefecture
  - Novartis Investigative Site, Kawachi-Nagano, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Fuchū, Tokyo
  - Novartis Investigative Site, Ōme, Tokyo
  - Novartis Investigative Site, Shimonoseki, Yamaguchi
  - Novartis Investigative Site, Chūō, Yamanashi
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka
- Novartis Investigative Site, Beirut, Lebanon
- Novartis Investigative Site, Guadalajara, Jalisco, Mexico
- Netherlands (3):
  - Novartis Investigative Site, Almelo, Overijssel
  - Novartis Investigative Site, Rotterdam, South Holland
  - Novartis Investigative Site, Groningen
- Poland (3):
  - Novartis Investigative Site, Bytom
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
- South Africa (2):
  - Novartis Investigative Site, Cape Town, Western Cape
  - Novartis Investigative Site, Stellenbosch, Western Cape
- Spain (7):
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Bilbao, Bizkaia
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Stockholm, SE, Sweden
- Switzerland (3):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Fribourg
  - Novartis Investigative Site, Sankt Gallen
- United Kingdom (3):
  - Novartis Investigative Site, Barnet
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Sun MM, Pope JE. Polymyalgia rheumatica and giant cell arteritis: diagnosis and management. Curr Opin Rheumatol. 2025 Jan 1;37(1):32-38. doi: 10.1097/BOR.0000000000001059. Epub 2024 Oct 14. PMID 39400109